CLINICAL TRIAL: NCT06556277
Title: Acute Consequences of Glucocorticoid Secretion in Overweight and Obese Individuals During Maximum Calorie Intake: a Double-blind, Randomized, Placebo-controlled, Cross-over Study
Brief Title: Acute Consequences of Glucocorticoid Secretion in Overweight and Obese Individuals During Maximum Calorie Intake
Acronym: Gluco-Max
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eleonora Seelig (Other)
Responsible Party: Sponsor-Investigator, Eleonora Seelig, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EKNZ 2024-01381
Record Dates: First submitted 2024-07-17; First posted 2024-08-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Glucocorticoids; Overweight and Obesity; Overeating
MeSH Terms: conditions — Overweight; Obesity; Hyperphagia | interventions — Metyrapone; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled cross-over study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metyrapone And Hydrocortisone (Experimental): During one of the study periods, subjects receive hydrocortisone 19.9 mg/d day 1 to day 6 and 12 mg/d on day 7 subcutaneously via a pump in a pulsed fashion (eight times/day) and metyrapone per os (starting with a dose of 750 mg/d, then the dose will be increased on day 3, where 2500mg/d is achieved and reduced on day 7 to 750mg).
  Interventions: Drug: Metyrapone And Hydrocortisone
- Placebo (Placebo Comparator): During the other study period, subjects receive placebo (0,9% NaCl solution) the same dose of placebo instead of hydrocortisone subcutaneously via a pump in a pulsed fashion and the same dose of placebo tablets p.o instead of metyrapone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metyrapone And Hydrocortisone — Drug: Metyrapone 250 mg Oral Tablets
  During one phase of the study: Metyrapone (pills of 250mg) on full stomach: Day 1 0-1-2, day 2 1-2-2, day 3 3-3-4 day 4 3-3-4 day 5 3-3-4 day 6 3-3-4 day 7 3-0-0
  Drug: Hydrocortisone 19,9mg/12mg s.c., pulsatile with a flow rate of 10μl/s
  Hydrocortisone will be delivered subcutaneously via a pump in a pulsed fashion with a flow rate of 10μl/s from day 1 to day 6 in a total daily dose of 19.9mg and 12mg on day 7
  Arms: Metyrapone And Hydrocortisone
Drug: Placebo — Drug: Placebo 250 mg Tablets
  During another phase of the study: identical looking placebo pills starting Day 1 During one phase of the study: Metyrapone (pills of 250mg) on full stomach: Day 1 0-1-2, day 2 1-2-2, day 3 3-3-4 day 4 3-3-4 day 5 3-3-4 day 6 3-3-4 day 7 3-0-0
  Drug: Placebo (0,9% NaCl solution)
  Placebo (0,9% NaCl solution) 19.9 mg/d subcutaneously via a pump in a pulsed fashion with a flow rate of 10μl/s from day 1 to day 6 and 12mg on day 7
  Arms: Placebo

SUMMARY:
The investigator aim to understand whether food-induced glucocorticoids influence fat mass in overweight and obese people.

In a randomized, cross-over study, 23 overweight and obese volunteers will receive a block and replace therapy that mimics physiological glucocorticoid (GC) rhythm (metyrapone plus hydrocortisone) or placebo. Participants will undergo two identical overfeeding periods with each treatment. With the block and replace therapy food-induced GC peak will be suppressed. Metabolic and immunological parameters will be compared to reveal the effects of GCs during excessive overfeeding, particularly to understand changes in body fat.

DETAILED DESCRIPTION:
Obesity is one of the most serious health problems of the 21st century, and new therapies are urgently needed.

Glucocorticoids (GCs) increase with acute food intake. Several clinical studies have found that glucocorticoids contribute to common obesity, but the underlying mechanisms remain unknown. Here, the investigator aim to understand whether GCs influence the total body fat in obese and overweight study participants during excessive overfeeding.

In a randomized, cross-over study, 23 overweight and obese individuals will receive a block and replace therapy that mimics physiological GC rhythm (Metyrapone plus hydrocortisone) or placebo. Participants will undergo two identical overfeeding periods with each treatment. With the block and replace therapy, food-induced GC peak will be suppressed. Metabolic, autonomic, and immunological parameters will be compared.

A) Participants will receive hydrocortisone 19.9mg/d day 1 to day 6 and 12mg on day 7 subcutaneously via a pump in a pulsed fashion (eight times/day) and metyrapone per os (starting with a dose of 750mg/d on day 1 to 2500mg on day 3, which will be kept constant until day 6 and then reduced to 750mg on day 7)

B) Participants will receive placebo (0,9% NaCl solution) 19.9mg/d day 1 to day 6 and 12mg on day 7 subcutaneously via a pump in a pulsed fashion (eight times/day) and placebo pills per os (starting with a dose of 750mg/d on day 1 to 2500mg on day 3, which will be kept constant until day 6 and then reduced to 750mg on day 7)

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 to 50 years
* BMI≥ 25 kg/m² with a stable weight within past three months before study initiation

Exclusion Criteria:

* Any severe acute or chronic disease, including diabetes mellitus type 2
* Intake of GLP-1 agonists or hormone therapy
* Hypercortisolism
* Casual smoking (more than 6 cigarettes per day)
* Frequent, heavy alcohol consumption (more than 30g/day)
* Frequent, heavy caffeine consumption (more than 4 caffeinated drinks/day)
* Regular physical exercise (more than 4hrs per week)
* Shift work
* Participation in an investigational drug trial within the past two months
* Intake of any steroid-containing drugs, including topical steroids and inhalers, within 4 weeks of the study initiation
* Known allergy to metyrapone
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since hormone fluctuations associated with the menstrual cycle may alter cortisol levels, women will not be included in the study. Although diversity will be reduced and the statements of the study cannot be applied to the female sex, these strict inclusion criteria allow an optimal homogeneity and increase statistical power.
Enrollment: 23 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Total body fat | Two 7-day intervention periods
  Change in total body fat assessed with a Dual-Energy-X-Ray-Absorptiometry (DXA)

SECONDARY OUTCOMES:
Total lean mass | Two 7-day intervention periods
  Change in total lean mass assessed with DXA
Insulin sensitivity | Two 7-day intervention periods
  Change in insulin sensitivity assessed with a mixed meal tolerance test
Glucose | Two 7-day intervention periods
  Change in Glucose assessed with a mixed meal tolerance test
Insulin | Two 7-day intervention periods
  Change in Insulin assessed with a mixed meal tolerance test
C-peptide | Two 7-day intervention periods
  Change in C-peptide assessed with a mixed meal tolerance test
Energy expenditure | Two 7-day intervention periods
  Basal metabolic rate measured with indirect calorimetryy
Substrate utilization | Two 7-day intervention periods
  Respiratory quotient assessed with indirect calorimetry
Systolic and diastolic blood pressure | Two 7-day intervention periods
  Assessment of blood pressure with a standard blood pressure monitor.
Weight | Two 7-day intervention periods
  Measurement of weight with a standard scale
Lipids (mmol/l) ((total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides) | Two 7-day intervention periods
  Blood sample
Immune cells (peripheral blood mononuclear cells) | Two 7-day intervention periods
  Blood sample
Satiation | Two 7-day intervention periods
  Amount of food intake with ad libitum buffet
Satiety | Two 7-day intervention periods
  Appetite rating with visual analogue scale (VAS) from 0mm-100mm (0mm=not at all and 100mm=extreme)
Motivation | Two 7-day intervention periods
  Motivation to eat measured with a speed clicking test
IL-6 (Inflammatory markers) | Two 7-day intervention periods
  Blood sample
IL-1RA (Inflammatory markers) | Two 7-day intervention periods
  Blood sample
IL-8 (Inflammatory markers) | Two 7-day intervention periods
  Blood sample
CRP (Inflammatory markers) | Two 7-day intervention periods
  Blood sample
Thyroid hormones | Two 7-day intervention periods
  Blood sample
Growth hormone | Two 7-day intervention periods
  Blood sample
IGF1 | Two 7-day intervention periods
  Blood sample
Catecholamines | Two 7-day intervention periods
  Blood sample
GLP-1 | Two 7-day intervention periods
  Blood sample
GIP | Two 7-day intervention periods
  Blood sample
Glucagon | Two 7-day intervention periods
  Blood sample
PYY | Two 7-day intervention periods
  Blood sample
CCK | Two 7-day intervention periods
  Blood sample
FGF21 | Two 7-day intervention periods
  Blood sample
Leptin | Two 7-day intervention periods
  Blood sample
Ghrelin | Two 7-day intervention periods
  Blood sample
GDF15 | Two 7-day intervention periods
  Blood sample
Cortisol | Two 7-day intervention periods
  Blood sample
Aldosterone | Two 7-day intervention periods
  Blood sample
Renin | Two 7-day intervention periods
  Blood sample
ACTH | Two 7-day intervention periods
  Blood sample
Pregnenolone | Two 7-day intervention periods
  Blood sample
Progesterone | Two 7-day intervention periods
  Blood sample
11-deoxycorticosterone | Two 7-day intervention periods
  Blood sample
Corticosterone | Two 7-day intervention periods
  Blood sample
18-hydroxycorticosterone | Two 7-day intervention periods
  Blood sample
17-hydroxypregnenolone | Two 7-day intervention periods
  Blood sample
17-hydroxyprogesterone | Two 7-day intervention periods
  Blood sample
11-deoxycortisol | Two 7-day intervention periods
  Blood sample
Oxytocin | Two 7-day intervention periods
  Blood sample

OTHER OUTCOMES:
Untargeted metabolomics of blood | Two 7-day intervention periods
  Blood sample
Untargeted metabolomics of adipose tissue | Two 7-day intervention periods
  Adipose tissue sample
Untargeted metabolomics of muscle | Two 7-day intervention periods
  Muscle tissue sample
Gene expression analysis of adipose tissue | Two 7-day intervention periods
  Adipose tissue sample
Gene expressions analysis of muscle tissue | Two 7-day intervention periods
  Muscle tissue sample

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Seelig, PD Dr.med., Principal Investigator — Sponsor and principal investigator
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No